CLINICAL TRIAL: NCT02985515
Title: Steroid Nasal Irrigation for Flavor Evaluation and Detection (SNIFFED) Study
Brief Title: Steroid Nasal Irrigation for Flavor Evaluation and Detection Study
Acronym: SNIFFED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201608163
Record Dates: First submitted 2016-12-03; First posted 2016-12-07 (Estimated); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Olfactory Disorder
Keywords: Anosmia; Hyposmia; Intranasal Steroid Irrigation; Olfactory Neuroplasticity; Olfactory training
MeSH Terms: conditions — Anosmia | interventions — Olfactory Training

STUDY DESIGN:
Intervention Model Description: This is a prospective cohort, pre- and post-intervention study
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Budesonide Nasal Irrigation (No Intervention): 30-day run-in course of budesonide nasal irrigation.
  1-month supply of budesonide capsules, an 8-oz sinus rinse bottle, and a 1-month supply of commercially prepared isotonic salt packets.
  Participants were instructed to dissolve 2 budesonide capsules (0.5mg per capsule) into the sinus rinse bottle along with the saline mixture and then irrigate both nasal cavities once daily.
- Budesonide Nasal Irrigation + Smell Training (Experimental): Budesonide nasal irrigation + smell training for 12 weeks
  Interventions: Behavioral: Smell training
- Controls (No Intervention): Baseline olfaction testing and rs-fMRI

INTERVENTIONS:
Behavioral: Smell training — Participants will be provided with 4 vials of essential odors. Participants will sniff each scent for 20-30 seconds, twice daily, for 12 weeks. The participant will take 30 seconds of rest between each scent. All participants will undergo this smell training regimen for 12 weeks.
  Other Names: Olfactory Training
  Arms: Budesonide Nasal Irrigation + Smell Training

SUMMARY:
The purpose of this research study is to examine the efficacy of a 12-week smell training intervention for participants with olfactory dysfunction following an infection of the upper respiratory tract.

DETAILED DESCRIPTION:
Olfactory dysfunction affects up to fifteen percent of the general population and can cause significant psychosocial distress including decreased appetite, reduced self-hygiene, and mood disturbances.

This study aims to study the efficacy of smell training for patients with olfactory dysfunction following a viral upper respiratory tract infection. Eligible participants will complete a 30-day course of budesonide nasal saline irrigation. Participants who do not show improvement in their olfaction based on composite smell and taste tests will be eligible to receive a baseline resting-state fMRI (rs-fMRI) and complete a 12-week smell training intervention program. Smell training involves participants smelling 4 odors (phenyl ethyl alcohol, eucalyptus, lemon, and eugenol) twice a day for 12 weeks. Following completion of smell training, participants will undergo repeat smell and taste tests as well as rs-fMRI to ascertain the efficacy of smell training.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* Anosmia or hyposmia (UPSIT <34 (male), UPSIT <34 (female); Sniffin' Sticks threshold below 5.5)

Exclusion Criteria:

* Inability to understand English
* Current smoker or history of smoking within the past 6 months
* Current nasal polyps
* Exposure to head and or/neck radiation
* Exposure to chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] Deems DA, Doty RL, Settle RG, Moore-Gillon V, Shaman P, Mester AF, Kimmelman CP, Brightman VJ, Snow JB Jr. Smell and taste disorders, a study of 750 patients from the University of Pennsylvania Smell and Taste Center. Arch Otolaryngol Head Neck Surg. 1991 May;117(5):519-28. doi: 10.1001/archotol.1991.01870170065015. PMID 2021470
- [Background] Doty RL, Frye RE, Agrawal U. Internal consistency reliability of the fractionated and whole University of Pennsylvania Smell Identification Test. Percept Psychophys. 1989 May;45(5):381-4. doi: 10.3758/bf03210709. PMID 2726398
- [Background] Hummel T, Sekinger B, Wolf SR, Pauli E, Kobal G. 'Sniffin' sticks': olfactory performance assessed by the combined testing of odor identification, odor discrimination and olfactory threshold. Chem Senses. 1997 Feb;22(1):39-52. doi: 10.1093/chemse/22.1.39. PMID 9056084
- [Background] Kobal G, Hummel T, Sekinger B, Barz S, Roscher S, Wolf S. "Sniffin' sticks": screening of olfactory performance. Rhinology. 1996 Dec;34(4):222-6. PMID 9050101
- [Background] Coldwell SE, Mennella JA, Duffy VB, Pelchat ML, Griffith JW, Smutzer G, Cowart BJ, Breslin PA, Bartoshuk LM, Hastings L, Victorson D, Hoffman HJ. Gustation assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S20-4. doi: 10.1212/WNL.0b013e3182872e38. PMID 23479539
- [Background] Bartoshuk LM, Duffy VB, Hayes JE, Moskowitz HR, Snyder DJ. Psychophysics of sweet and fat perception in obesity: problems, solutions and new perspectives. Philos Trans R Soc Lond B Biol Sci. 2006 Jul 29;361(1471):1137-48. doi: 10.1098/rstb.2006.1853. PMID 16815797
- [Background] Pepino MY, Finkbeiner S, Beauchamp GK, Mennella JA. Obese women have lower monosodium glutamate taste sensitivity and prefer higher concentrations than do normal-weight women. Obesity (Silver Spring). 2010 May;18(5):959-65. doi: 10.1038/oby.2009.493. Epub 2010 Jan 14. PMID 20075854
- [Background] Cicerale S, Breslin PA, Beauchamp GK, Keast RS. Sensory characterization of the irritant properties of oleocanthal, a natural anti-inflammatory agent in extra virgin olive oils. Chem Senses. 2009 May;34(4):333-9. doi: 10.1093/chemse/bjp006. Epub 2009 Mar 8. PMID 19273462
- [Background] Keast RS, Roper J. A complex relationship among chemical concentration, detection threshold, and suprathreshold intensity of bitter compounds. Chem Senses. 2007 Mar;32(3):245-53. doi: 10.1093/chemse/bjl052. Epub 2007 Jan 13. PMID 17220518
- [Background] Cowart BJ. Relationships between taste and smell across the adult life span. Ann N Y Acad Sci. 1989;561:39-55. doi: 10.1111/j.1749-6632.1989.tb20968.x. No abstract available. PMID 2735688
- [Background] Hummel T, Rissom K, Reden J, Hahner A, Weidenbecher M, Huttenbrink KB. Effects of olfactory training in patients with olfactory loss. Laryngoscope. 2009 Mar;119(3):496-9. doi: 10.1002/lary.20101. PMID 19235739
- [Background] Stamps JJ, Bartoshuk LM, Heilman KM. A brief olfactory test for Alzheimer's disease. J Neurol Sci. 2013 Oct 15;333(1-2):19-24. doi: 10.1016/j.jns.2013.06.033. Epub 2013 Aug 5. PMID 23927938
- [Background] Tepper BJ, Christensen CM, Cao J. Development of brief methods to classify individuals by PROP taster status. Physiol Behav. 2001 Jul;73(4):571-7. doi: 10.1016/s0031-9384(01)00500-5. PMID 11495661
- [Background] Pekala K, Chandra RK, Turner JH. Efficacy of olfactory training in patients with olfactory loss: a systematic review and meta-analysis. Int Forum Allergy Rhinol. 2016 Mar;6(3):299-307. doi: 10.1002/alr.21669. Epub 2015 Dec 1. PMID 26624966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults 18 to 70 years of age with clinically diagnosed or self reported postviral olfactory loss of 3 months or longer were eligible to participate.
  For the control group, adults with normal smell function were eligible to participate.
Pre-assignment Details: PVOD participants first underwent 30-day trial period of budesonide nasal irrigation. If they did not experience improvement in their smell to the normal range as measured by UPSIT and Sniffin'Sticks, they continued budesonide nasal irrigation plus 12-weeks of smell intervention. Resting-state fMRI was obtained before and after smell intervention.
  For the participants in the Control Group, one time fs-MRI and questionnaire completion only.
Groups:
- Controls: Healthy volunteers with normal smell function. Participants in the Control Group completed UPSIT, MRI, and Questionnaires one time and were finished with study participation.
Period: Olfaction Testing
Arm/Group | Controls | Budesonide Nasal Irrigation
Started (30 day period) | 20 | 31
Completed | 20 | 23
Not Completed | 0 | 8
Not completed — Lost to Follow-up | 0 | 5
Not completed — Protocol Violation | 0 | 3
Period: Smell Training
Arm/Group | Controls | Budesonide Nasal Irrigation
Started | 0 | 23
Completed | 0 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data were only *collected* for 23 participants in the Budesonide Nasal Irrigation Arm/Group
Groups:
- Budesonide Nasal Irrigation: Participants will first undergo a 30-day trial of budesonide nasal saline irrigation. If there is no subsequent improvement in olfaction, participants will undergo a 12-week smell training intervention.
  Budesonide nasal irrigation: Eligible participants will be provided with a "NeilMed" Sinus Rinse Regular Bottle Kit and a one-month supply of USP Grade Sodium Chloride & Sodium Bicarbonate Mixture commercially prepared packets. Participants will need to purchase distilled water or boil tap water for five minutes for use with the saline irrigation. The contents of two capsules (0.5mg budesonide each) will be dissolved into "NeilMed" Sinus Rinse Regular Bottle along with the saline rinse. Both nasal cavities will be irrigated once daily for 30 days.
  Smell training: Participants who do not have objective improvement in their olfaction after the trial of budesonide irrigation will have a baseline resting-state fMRI (rs-fMRI) and undergo 12 weeks of smell training. Smell training involves the participants smelling 4 vials of essential odors (clove, lemon, eucalyptus, rose) twice a day for 12 weeks. Following smell training, participants will have their smell ability re-evaluated and a second rs-fMRI performed.
- Control Group: Control participants sex and age matched (±5 years) to participants with PVOD had normal smell as determined by UPSIT and were recruited for baseline neuroimaging. Individuals with MRI contraindications were excluded.
- Total: Total of all reporting groups
Arm/Group | Budesonide Nasal Irrigation | Control Group | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Categorical [Count of Participants; unit: Participants] — Population: A total of 31 PVOD participants were in the Budesonide Nasal Irrigation group. Of the 31 participants, 23 participants remained after 8 were removed for protocol violations. The remaining 23 participants showed no improvement after the 30 days of budesonide nasal irrigation and therefore continued on the study and received 12 weeks of smell training.
  20 participants in the Control Group.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 15 | 20 | 35
    >=65 years | 8 | 0 | 8
Age, Continuous [Median (Full Range); unit: years] — Population: A total of 31 PVOD participants were in the Budesonide Nasal Irrigation group. Of the 31 participants, 23 remained after 8 were removed for protocol violations. The remaining 23 showed no improvement after the 30 days of budesonide nasal irrigation and therefore continued on the study and received 12 weeks of smell training. Additionally, 7 participants were removed from the final analysis due to motion artifact on MRI leaving a total of 16 participants in the final analysis.
  years | 62 [30 to 70] | 61.5 [30 to 69] | 62 [30 to 70]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total of 31 PVOD participants were in the Budesonide Nasal Irrigation group. Of the 31 participants, 23 remained after 8 were removed for protocol violations. The remaining 23 showed no improvement after the 30 days of budesonide nasal irrigation and therefore continued on the study and received 12 weeks of smell training. Additionally, 7 participants were removed from the final analysis due to motion artifact on MRI leaving a total of 16 participants in the final analysis.
  Participants
    Female | 17 | 15 | 32
    Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 31 PVOD participants were in the Budesonide Nasal Irrigation group. Of the 31 participants, 23 remained after 8 were removed for protocol violations. The remaining 23 showed no improvement after the 30 days of budesonide nasal irrigation and therefore continued on the study and received 12 weeks of smell training. Additionally, 7 participants were removed from the final analysis due to motion artifact on MRI leaving a total of 16 participants in the final analysis.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 2 | 4
    White | 21 | 18 | 39
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: A total of 31 PVOD participants were in the Budesonide Nasal Irrigation group. Of the 31 participants, 23 remained after 8 were removed for protocol violations. The remaining 23 showed no improvement after the 30 days of budesonide nasal irrigation and therefore continued on the study and received 12 weeks of smell training. Additionally, 7 participants were removed from the final analysis due to motion artifact on MRI leaving a total of 16 participants in the final analysis.
  Participants
    United States | 23 | 20 | 43
Duration of smell loss [Median (Full Range); unit: months] — Baseline duration of smell loss was not obtained from the control group as all 20 participants in the control group had normal smell. Population: A total of 31 PVOD participants were in the Budesonide Nasal Irrigation group. Of the 31 participants, 23 remained after 8 were removed for protocol violations. The remaining 23 showed no improvement after the 30 days of budesonide nasal irrigation and therefore continued on the study and received 12 weeks of smell training. Data were only *collected* for 23 participants in the Budesonide Nasal Irrigation Arm/Group
  months
    number analyzed (Participants) | 23 | 0 | 23
    (all) | 12 [3 to 240] |  | 12 [3 to 240]
UPSIT [Median (Full Range); unit: units on a scale] — University of Pennsylvania Identification Test (UPSIT) consists of 4 odor-impregnated booklets that participants scratch and sniff to identify various odors, and scores account for differences in sex. Hyposmia is defined as a score of 19 to 34 for females and 19 to 33 for males. Anosmia for either sex is defined as a score below 18. A score below 5 is highly suggestive of malingering. Possible scores range from 0 to 40 with higher scores indicating better sense of smell. Population: A total of 31 PVOD participants were in the Budesonide Nasal Irrigation group. Of the 31 participants, 23 remained after 8 were removed for protocol violations. The remaining 23 showed no improvement after the 30 days of budesonide nasal irrigation and therefore continued on the study and received 12 weeks of smell training. Data were only *collected* for 23 participants in the Budesonide Nasal Irrigation Arm/Group
  units on a scale
    number analyzed (Participants) | 23 | 0 | 23
    (all) | 19.5 [7 to 36] |  | 35 [10 to 39]
TDI [Median (Full Range); unit: units on a scale] — Like UPSIT, the Sniffin' Sticks test is a reliable and validated tool to assess olfactory function. Sniffin' Sticks are odor-encapsulated markers that are used to measure odor detection threshold, discrimination, and identification (TDI). Normosmia is defined as a TDI score >30.5. An increase by 5.5 points or more from baseline is considered meaningful improvement. Possible scores range from 1 to 48 with higher values indicating better sense of smell.
  Baseline TDI was not obtained from the control group as all 20 participants had normal smell. Population: A total of 31 PVOD participants were in the Budesonide Nasal Irrigation group. Of the 31 participants, 23 remained after 8 were removed for protocol violations. The remaining 23 showed no improvement after the 30 days of budesonide nasal irrigation and therefore continued on the study and received 12 weeks of smell training. Data were only *collected* for 23 participants in the Budesonide Nasal Irrigation Arm/Group
  units on a scale
    number analyzed (Participants) | 23 | 0 | 23
    (all) | 18 [7 to 30.5] |  | 18 [7 to 30.5]
VAS sense of smell [Median (Full Range); unit: units on a scale] — Baseline subjective sense of smell was measured using visual analogue sense of smell with scores ranging from 0 to 100. 0 represented no sense of smell and 100 represented best possible sense of smell.
  As all participants in the control group had normal sense of smell, baseline VAS was not measured. Population: A total of 31 PVOD participants were in the Budesonide Nasal Irrigation group. Of the 31 participants, 23 remained after 8 were removed for protocol violations. The remaining 23 showed no improvement after the 30 days of budesonide nasal irrigation and therefore continued on the study and received 12 weeks of smell training. Data were only *collected* for 23 participants in the Budesonide Nasal Irrigation Arm/Group.
  units on a scale
    number analyzed (Participants) | 23 | 0 | 23
    (all) | 0.1095 [0 to 0.5] |  | 0.1095 [0 to 0.5]
QOD-NS score [Median (Full Range); unit: units on a scale] — The Questionnaire for Olfactory Dysfunction-Negative Statements (QOD-NS) is a validated 17-item questionnaire that pertains to olfactory-specific quality of life domains adversely impacted by olfactory dysfunction and is inversely scored (scores range from 0 to 51), with higher scores reflective of more impaired quality of life.
  As all participants in the control group had both objective and subjective normal sense of smell, QOD-NS was not ascertained in the control group. Population: A total of 31 PVOD participants were in the Budesonide Nasal Irrigation group. Of the 31 participants, 23 remained after 8 were removed for protocol violations. The remaining 23 showed no improvement after the 30 days of budesonide nasal irrigation and therefore continued on the study and received 12 weeks of smell training. Data were only *collected* for 23 participants in the Budesonide Nasal Irrigation Arm/Group.
  units on a scale
    number analyzed (Participants) | 23 | 0 | 23
    (all) | 10.55 [3.42 to 16.53] |  | 10.55 [3.42 to 16.53]

OUTCOME MEASURES:

1. Primary Outcome: Pre- and Post-intervention Difference in Functional Connectivity Before and After Smell Training.
Description: Baseline and post-intervention connectivity within and between regions of interest in the olfactory and olfactory related networks using resting state fMRI will be obtained. Resting-state connectivity was analyzed using the CONN toolbox version 18b (https://web.conn-toolbox.org/) and SPM12, version 7487 (Wellcome Trust Centre for Neuroimaging). Functional connectivity values (Fisher z-transformed Pearson correlation coefficients) were compared using a paired, 2-tailed t test and corrected for multiple comparisons. p<0.05 was considered to be significant.
Time Frame: 12 weeks
Population: Of the total 23 participants who completed smell training and rs-fMRI, 7 were excluded from analysis because of excessive artifact. Thus, the final study included a total of 16 participants. A set of 164 regions of interest(ROIs) from the CONN toolbox were used, supplemented with 23 ROIs determined by prior studies to be associated with olfactory processing. The CONN toolbox is an open source Matlab/SPM software that integrates pre-processing, display, and analysis of rs-fMRI data.
Measure: Number; unit: Regions of interest
Units Other Than Participants: Regions of interest
Groups:
- Smell Training: Participants will first undergo a 30-day trial of budesonide nasal saline irrigation. If there is no subsequent improvement in olfaction, participants will undergo a 12-week smell training intervention.
  Smell training: Eligible participants will be provided with a "NeilMed" Sinus Rinse Regular Bottle Kit and a one-month supply of USP Grade Sodium Chloride & Sodium Bicarbonate Mixture commercially prepared packets. Participants will need to purchase distilled water or boil tap water for five minutes for use with the saline irrigation. The contents of two capsules (0.5mg budesonide each) will be dissolved into "NeilMed" Sinus Rinse Regular Bottle along with the saline rinse. Both nasal cavities will be irrigated once daily for 30 days.
  Participants who do not have objective improvement in their olfaction after the trial of budesonide irrigation will have a baseline resting-state fMRI (rs-fMRI) and undergo 12 weeks of smell training. Smell training involves the participants smelling 4 vials of essential odors twice a day for 12 weeks. Following smell training, participants will have their smell ability re-evaluated and a second rs-fMRI performed.
Arm/Group | Smell Training
Number analyzed (Participants) | 16
Number analyzed (Regions of interest) | 187
Regions of interest | 5

2. Secondary Outcome: Pre- and Post-intervention Difference in Smell Testing Before and After Budesonide Treatment
Description: Objective pre- and post-intervention differences of participant performance on the UPSIT and Sniffin Sticks tests before and after budesonide saline nasal irrigation.
  University of Pennsylvania Identification Test (UPSIT) consists of 4 odor-impregnated booklets that participants scratch and sniff to identify various odors, and scores account for differences in sex. Hyposmia is defined as a score of 19 to 34 for females and 19 to 33 for males. Anosmia for either sex is defined as a score below 18. Possible scores range from 0 to 40 with higher scores indicating better sense of smell.
  Sniffin' Sticks are odor-encapsulated markers that are used to measure odor detection threshold, discrimination, and identification (TDI). Normosmia is defined as a TDI score >30.5. An increase by 5.5 points or more from baseline is considered meaningful improvement. Possible scores range from 1 to 48 with higher values indicating better sense of smell.
Time Frame: 30 days
Measure: Median (Full Range); unit: units on a scale
Groups:
- Budesonide Nasal Irrigation: Participants will first undergo a 30-day trial of budesonide nasal saline irrigation. If there is no subsequent improvement in olfaction, participants will undergo a 12-week smell training intervention.
  Budesonide nasal irrigation: Eligible participants will be provided with a "NeilMed" Sinus Rinse Regular Bottle Kit and a one-month supply of USP Grade Sodium Chloride & Sodium Bicarbonate Mixture commercially prepared packets. Participants will need to purchase distilled water or boil tap water for five minutes for use with the saline irrigation. The contents of two capsules (0.5mg budesonide each) will be dissolved into "NeilMed" Sinus Rinse Regular Bottle along with the saline rinse. Both nasal cavities will be irrigated once daily for 30 days.
Arm/Group | Budesonide Nasal Irrigation
Number analyzed (Participants) | 16
units on a scale
  UPSIT | 19.5 [5 to 40]
  TDI | 17.5 [7 to 27.2]

3. Secondary Outcome: Subjective Response to Smell Training Intervention
Description: Participants subjective sense of smell following intervention is measured using a visual analogue scale from 0 to 100 with 0 representing no sense of smell and 100 representing best possible sense of smell.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: units on a scale
Groups:
- Smell Training: Smell training: Participants had no improvement in olfaction underoing 30-days of budesonide nasal saline irrigation underwent 12-week smell training intervention. Participants were given 4 vials of essential oils (clove, lemon, eucalyptus, rose) to smell twice a day for 12 weeks. Participants underwent a baseline resting-state (rs-fMRI) prior to smell intervention. Following smell training, participants had their smell ability re-evaluated and a second rs-fMRI performed.
Arm/Group | Smell Training
Number analyzed (Participants) | 16
units on a scale | 23.8 [9 to 83.8]

4. Secondary Outcome: Comparison of Olfactory Network in Healthy Controls to Study Participants
Description: Baseline functional connectivity within and between the olfactory and associated networks of healthy controls will be compared to that of study participants prior to smell intervention treatment as measured by rs-fMRI.Resting-state connectivity was analyzed using the CONN toolbox version 18b (https://web.conn-toolbox.org/) and SPM12, version 7487 (Wellcome Trust Centre for Neuroimaging). Functional connectivity values (Fisher z-transformed Pearson correlation coefficients) were compared using a paired, 2-tailed t test and corrected for multiple comparisons . P < .05 was considered statistically significant.
Time Frame: 1 week
Population: A set of 164 regions of interest (ROIs) from the CONN toolbox were used, supplemented with 23 ROIs determined by prior studies to be associated with olfactory processing.
Measure: Number; unit: Regions of interest
Units Other Than Participants: Regions of interest
Groups:
- Control Group: 20 participants sex and age matched (+/- 5 years) to participants with PVOD with normal smell as determined by UPSIT were recruited for baseline neuroimaging.
Arm/Group | Control Group
Number analyzed (Participants) | 20
Number analyzed (Regions of interest) | 187
Regions of interest | 13

5. Secondary Outcome: Pre- and Post-intervention Difference in Smell Testing Before and After Smell Training
Description: Objective pre- and post-intervention differences of participant performance on the UPSIT and Sniffin Sticks tests before and after budesonide saline nasal irrigation.
  University of Pennsylvania Identification Test (UPSIT) consists of 4 odor-impregnated booklets that participants scratch and sniff to identify various odors, and scores account for differences in sex. Hyposmia is defined as a score of 19 to 34 for females and 19 to 33 for males. Anosmia for either sex is defined as a score below 18. Possible scores range from 0 to 40 with higher scores representing better sense of smell.
  Sniffin' Sticks are odor-encapsulated markers that are used to measure odor detection threshold, discrimination, and identification (TDI). Normosmia is defined as a TDI score >30.5. An increase by 5.5 points or more from baseline is considered meaningful improvement. Possible scores range from 1 to 48 with higher values indicating better sense of smell.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: units on a scale
Groups:
- Smell Training: Smell training:
  Participants who do not have objective improvement in their olfaction after the trial of budesonide irrigation will have a baseline resting-state fMRI (rs-fMRI) and undergo 12 weeks of smell training. Smell training involves the participants smelling 4 vials of essential odors (clove, lemon, eucalyptus, rose) twice a day for 12 weeks. Following smell training, participants will have their smell ability re-evaluated and a second rs-fMRI performed.
Arm/Group | Smell Training
Number analyzed (Participants) | 16
units on a scale
  UPSIT | 19 [9 to 40]
  TDI | 18.3 [7 to 34.5]

6. Secondary Outcome: Pre and Post Difference in QOD-NS After Smell Training
Description: The QOD-NS is a validated 17-item questionnaire that pertains to olfactory-specific quality of life domains adversely impacted by olfactory dysfunction and is inversely scored (maximum score of 51), with higher scores reflective of more impaired quality of life.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Smell Training
Number analyzed (Participants) | 16
units on a scale | 7.4 [0 to 17.1]

ADVERSE EVENTS:
Time Frame: Up through 13 months
Description: # who underwent budesonide nasal irrigation at risk for serious adverse events:31; All participants who underwent the 12-weeks of smell training are included because all underwent 30-day trial of budesonide nasal irrigation. If improved, participation ended.If no improvement, they underwent 12-weeks of smell training intervention. # of controls at risk for serious adverse events:20; Adverse Events were not collected separately in the Smell Training portion from the Budesonide Nasal Irrigation.
Groups:
- Budesonide Nasal Irrigation: Adults 18 to 70 years of age with clinically diagnosed or self-reported postviral olfactory loss of 3 months underwent 30-day trial of budesonide nasal irrigation. If they improved, study participation ended. If they had no improvement in sense of smell after a 30-day trial of budesonide nasal irrigation, they then underwent 12-weeks of smell training intervention. All participants who underwent the 12-weeks of smell training intervention are included this adverse event group. Adverse Events were not collected separately in the Smell Training portion of the study from the Budesonide Nasal Irrigation but instead collected as a whole.
Arm/Group | Control Group | Budesonide Nasal Irrigation
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/31
Other Adverse Events (participants affected / at risk) | 3/20 | 2/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=20) | Budesonide Nasal Irrigation (N=31)
Cavernoma (Nervous system disorders) | 2 (2) | 0 (0) — Incidental MRI finding
pleomorphic adenoma (Nervous system disorders) | 1 (1) | 0 (0) — Incidental MRI finding
extra-axial meningiomas (Nervous system disorders) | 0 (0) | 2 (2) — Incidental MRI finding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT02985515/Prot_SAP_000.pdf